CLINICAL TRIAL: NCT02096432
Title: Suicide Prevention in Chinese Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Northwestern University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13110601; R34MH100443 (NIH)
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Behavioral: Behavioral Activation (Experimental): Behavioral Activation includes the following components: empowering education, referral to treatment, care Management, and behavior activation
  Interventions: Behavioral: Behavior Activation
- Usual Community Care (Other): Community standard care as usual
  Interventions: Behavioral: Usual Community Care

INTERVENTIONS:
Behavioral: Behavior Activation — Behavioral Activation includes the following components: empowering education, referral to treatment, care Management, and behavior activation
  Arms: Behavioral: Behavioral Activation
Behavioral: Usual Community Care — Community standard care as usual
  Arms: Usual Community Care

SUMMARY:
This project aims to develop and refine a suicide intervention protocol, and pilot test a culturally tailored randomized control trial to reduce suicidal thoughts among U.S. Chinese older adults. During the first phase of the study, the investigators plan to invite the community advisory board and key stakeholders to participate in the iterative design and refinement of the study protocol. During the second phase of the project and after the initial screening and based on a specific set of inclusion criteria, the investigators will invite U.S. Chinese older adult to participate in a pilot randomized control trial of a culturally adapted intervention to reduce the frequency and intensity of suicidal thoughts in Chinese older adults. During the third phase of the project, the investigators plan to invite pilot intervention participants as well as key stakeholders and health care professionals on the cultural acceptability of the pilot intervention. Through the achievement of these objectives, the investigators will set the foundation to fully test a culturally adapted in-home intervention, which may be particularly suitable for Chinese older adults with suicidal thoughts as it addresses cultural-specific barriers and integrates care management within existing community services agencies using non-mental health professionals, including community health workers.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as Chinese
2. >50 years of age
3. Suicidal thoughts within the last month as detected from the Item 9 in PHQ-9
4. No plans to move for 6 months
5. No significant cognitive impairment with Chinese Mini-Mental State Examination (C-MMSE) score >20

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-10; Primary Completion 2018-07 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Outcome measure will be measured in 10 weeks' time

CONTACTS AND LOCATIONS:
Overall Officials: XinQi Dong, MD, MPH, Principal Investigator — Rush University Medical Center; Melissa A. Simon, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Chinese community, Chicago, Illinois, United States